CLINICAL TRIAL: NCT06156540
Title: The Effect of Virtual Reality Glasses on the Psychological Well-Being and Care Burden of Patient Relatives Giving Care to Patients in the Palliative Care Clinic
Brief Title: Virtual Reality Glasses in Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Yadigar Ordu, Doctor Lecturer, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TUSEB
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Virtual Reality
Keywords: Virtual reality; Nursing; Palliative care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention was made to the control group. The posttest was administered four weeks after the pretest.As a result, caregivers' care burden and psychological well-being will be measured.
- Virtual Reality Group (Experimental): A pretest was administered to the experimental group. Then, 360-degree VR videos (nature walks, trips, etc.) were watched three days a week for four weeks. Then, the final test was administered.As a result, caregivers' care burden and psychological well-being will be measured.
  Interventions: Other: virtual reality glasses

INTERVENTIONS:
Other: virtual reality glasses — Using virtual reality glasses, caregivers in the experimental group were shown 360-degree VR relaxing videos.
  Arms: Virtual Reality Group

SUMMARY:
Developments in medicine and technology have led to an increase in life expectancy and an increase in the need for palliative care. palliative Care aims to reduce or eliminate a life-threatening situation. The palliative care team cares for the patient and provides informal support to the patient. It should provide care that centers on caregivers (patient's relatives). Relatives of patients who provide palliative care are responsible for their care As it increases, problems such as fatigue, hopelessness and anger may occur. Problems experienced by caregivers of patients Eliminating this problem and integrating it into care by providing psychosocial support is essential for the quality of care. caregivers Health technologies can be used to support In our research, we found that virtual reality glasses were used in palliative care clinics. It is aimed to investigate the effect of patient relatives who care for inpatients on the psychological well-being and care burden. A randomized controlled research design was used in the study. The population of the research is a country in Turkey between June and October 2023. The study consisted of patient relatives who provide care to patients in the palliative care clinic of the public hospital in the province. To research Relatives of patients who met the participation criteria and agreed to participate (control group, n=22; experimental group, n=22) constituted the sample. Data were collected from "Caregiver Introduction Form", "Psychological Well-Being Scale", "Caregiving Burden Scale" and "Virtual Reality Glasses". It was collected using the "Satisfaction Form". Before starting the research, a preliminary study was conducted with four patient relatives. of research In the implementation, firstly the preliminary application of the data collection tools was made. Then, the experimental group was given weekly Videos containing 360-degree images were watched using virtual reality glasses for 30 minutes for three days. In the control group No intervention was made. At the end of the research, the final application of the data collection tools was made. From research The data obtained was analyzed with the SPSS 22.0 package program.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* No vision, hearing or perception impairment that prevents communication,
* Not using glasses to wear VR glasses,
* No psychiatric disease,
* Absence of complaints such as migraine, vertigo, active nausea, vomiting, headache,
* Not having someone to help you care for your patient.

Exclusion Criteria:

* Wanting to leave the research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
psychological well-being | Four weeks after pretest
  The psychological well-being levels of caregivers will be evaluated using the psychological well-being scale.Psychological well-being scale (PIOS):
  It was developed by Diener et al. in 2009 and consists of eight items. The scale measuring socio-psychological well-being is a single-factor and 7-point Likert type (1 = Strongly disagree, 7 = Strongly agree). The lowest score that can be obtained from the scale is 8 and the highest score is 56. A high score from the scale indicates high psychological well-being.

SECONDARY OUTCOMES:
Determine maintenance burden | Four weeks after pretest
  Using the caregiving burden scale, caregivers' caregiving burden will be measured.
  Caregiving burden scale:
  The scale, developed by Zarit et al. in 1980 and adapted into Turkish by İnci and Erdem (2008), consists of 22 statements that determine the impact of caregiving on the individual's life. Scale items are generally related to the social and emotional domain and are of 4-point Likert type (0 = Never, 4 = Almost always). The lowest score that can be obtained from the scale is 0 and the highest score is 88. A high scale score indicates that the distress experienced is high (0-20 points = no care burden, 21-40 points = light care burden, 41-60 points = moderate care burden, 61-88 points = heavy care burden).

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data may be requested from the principal investigator upon reasonable request.

REFERENCES:
- [Derived] Ordu Y, Yilmaz S. The effect of using virtual reality goggles on psychological well-being and care burden of informal caregivers of patients hospitalized in a palliative care clinic. Eur J Oncol Nurs. 2024 Dec;73:102711. doi: 10.1016/j.ejon.2024.102711. Epub 2024 Oct 9. PMID 39406181